CLINICAL TRIAL: NCT04110028
Title: Shorter Recovery Time After Critical Illness
Brief Title: Nicotinamide Riboside in Hospitalized Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: ChromaDex, Inc. (Industry)
Responsible Party: Principal Investigator, Arne Vasli Lund Søraas, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2017/1334C
Record Dates: First submitted 2019-09-20; First posted 2019-10-01 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Inflammation; Acute Illness
Keywords: Nicotinamide riboside; NAD+; Epigenetics; Aging; PARP
MeSH Terms: conditions — Inflammation | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to placebo or nicotinamide riboside (NR) in increasing doses. The safety of each dose will be evaluated before commencing the next phase. In each phase nicotinamide or placebo will be administered.
  The patients will use NR for 90 days. When all patients have completed their NR treatment the study will be unblinded and the follow-up visits at one year later and further on will be unblinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The safety committee will have access to unblinded results during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Nicotinamide riboside 250 mg (Experimental): One capsule of 250 mg each morning for three months
  Interventions: Drug: Nicotinamide riboside
- Nicotinamide riboside 500 mg (Experimental): One capsule of 250 mg each morning and afternoon for three months
  Interventions: Drug: Nicotinamide riboside
- Nicotinamide riboside 1000 mg (Experimental): Two capsules of 250 mg each morning and afternoon for three months
  Interventions: Drug: Nicotinamide riboside
- Nicotinamide riboside 2000 mg (Experimental): Four capsules of 250 mg each morning and afternoon for three months
  Interventions: Drug: Nicotinamide riboside
- Placebo for 250 mg nicotinamide riboside (Placebo Comparator): One capsule each morning for three months
  Interventions: Drug: Placebo
- Placebo for 500 mg nicotinamide riboside (Placebo Comparator): One capsule each morning and afternoon for three months
  Interventions: Drug: Placebo
- Placebo for 1000 mg nicotinamide riboside (Placebo Comparator): Two capsules each morning and afternoon for three months
  Interventions: Drug: Placebo
- Placebo for 2000 mg nicotinamide riboside (Placebo Comparator): Four capsules each morning and afternoon for three months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotinamide riboside — Nicotinamide riboside in different doses
  Arms: Nicotinamide riboside 1000 mg; Nicotinamide riboside 2000 mg; Nicotinamide riboside 250 mg; Nicotinamide riboside 500 mg
Drug: Placebo — Placebo
  Arms: Placebo for 1000 mg nicotinamide riboside; Placebo for 2000 mg nicotinamide riboside; Placebo for 250 mg nicotinamide riboside; Placebo for 500 mg nicotinamide riboside

SUMMARY:
Patients will receive oral nicotinamide riboside or placebo and clinical and paraclinical outcome will be determined

DETAILED DESCRIPTION:
Patients experiencing acute illness will often have a prolonged recovery time. The cause of this is unknown, but certain factors, like age, duration, and graveness of the illness, is associated with prolonged recovery. In this study, we will investigate whether nicotinamide riboside can shorten the recovery phase and improve outcome after acute illness.

ELIGIBILITY:
Inclusion criteria:

1. Adults > 18 years old, admitted to hospital with tissue damage, can be included when they are considered medically stable though still expected to remain hospitalized for at least 7 more days (from inclusion).
2. Preferably: Previously included in the Janus Cohort or any other cohort or study with stored biological samples.

Exclusion Criteria:

1. Allergy to NR or ingredients in capsules or placebo.
2. Patients expected to pass away within 90 days.
3. Patients unable to give their consent
4. Unstable patients:

   i. Uncontrolled infection (clinical septicaemia, inadequate response to treatment, inadequate control of source of infection or at treating physician's discretion).

   ii. Mean arterial pressure <70 mm Hg and symptoms of hypotension. iii. Patients requiring dialysis at the time of inclusion or glomerular filtration rate <40 iv. Liver failure with Child-Pugh class B or C or any class associated with hepatic encephalopathy (any grade), alanin aminotransferase or aspartate aminotransferase >3 times upper limit v. Moderate to severe peripheral oedema and/or pulmonary oedema, any unstable cardiac rhythm, myocardial infarction with peak TNT >300 past week. Signs of elevated intracranial pressure (headache, vomiting and depressed global consciousness in conjunction with focal neurological signs, papilledema, spontaneous periorbital bruising and a triad of bradycardia, respiratory depression and hypertension).

   vi. Arterial pH <7.30 or >7.50 vii. Serum potassium under 3,2 or over 5 mmol/L.
5. Pregnancy or breastfeeding *
6. Any cancer not in full remission for >10 years
7. Use of St John's Wort based supplements during the past 30 days
8. Patient has undergone solid organ transplantation
9. Participation in any clinical trial with unknown medications
10. Major gastrointestinal or other internal bleeding past week
11. Logistical challenges after discharge. Patient must be able to attend follow up.
12. The treating physician considers the patient unfit or unable to participate. *All fertile women must have a human chorionic gonadotropin test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Length of stay from randomization to discharge from hospital to home or to an institution with a lower care level than a hospital for instance a long term care facility. | Up to 90 days
  Days

SECONDARY OUTCOMES:
Time to normalization of urine production | Up to 90 days
  Measured in ml/hour
Mortality | At 90 days, 65 weeks and 10 years
  Number of deaths
Length of stay from randomization to medically fit for discharge from hospital to home or to an institution with a lower care level than a hospital for instance a long term care facility. | Up to 90 days
  Days
Time to normalization of blood pressure | Up to 90 days
  Hours/days
Change in blood pressure during the study period | Baseline and 90 days and 65 weeks
  mmHg
Days on respiratory support | Up to 90 days
  Days
Number of days with temperature above 38 at any point from inclusion to discharge. | Up to 90 days
  Days
Number of days with temperature above 38 at any point from inclusion to discharge divided on number of days from inclusion to discharge | 90 days
  Number of days
Duration of stay in ICU after randomization | Up to 90 days
  Days
Number of newly diagnosed infections with identified agent from inclusion to end of trial | 90 days and 65 weeks
  Number
Number of newly diagnosed infections from inclusion to end of trial | 90 days and 65 weeks
  Number
Days on antibiotics from inclusion to end of trial | 90 days and 65 weeks
  Days
Days from inclusion to first antibiotic free day | Up to 90 days
  Days
Highest CRP from inclusion to end of trial | Up to 90 days
  CRP value
Changes in DNA methylation clocks | At baseline, 90 days and 65 weeks.
  Changes in the published DNA methylation clocks by Steve Horvath (Multi tissue, 2013, Skin and Blood, 2018, PhenoAge 2017, GrimAge 2018, telomere length 2019) and Hannum (Hannum clock 2013), Yan Zhang (continous Zhang score, 2017), AgeLab01 (Poster, Gordon Conference, Biology of Aging, July, 2019). All clocks are algorithms based on the Illumina "EPIC" DNA methylation BeadArray.
Changes in DNA methylation measured by the Illumina DNA methylation BeadArray | At baseline, 90 days and 65 weeks.
  Methylation sites (CpG sites) that are differentially changed in the intervention groups compared to the placebo group(s) over the studied time period. Correction for multiple testing will be done.
Change in quality of life | 14 days prior to admission, baseline, 90 days and 65 weeks
  EQ-5D-5L (Quality of life instrument developed by the EuroQol group). Scores ranging from 11111 (full health) to 33333/55555 (worst health).
Change in Katz activities of daily living | 14 days prior to admission, baseline, 90 days and 65 weeks
  Measured at pre-baseline (-14 days), 90 days and 65 weeks. Score 0-6 describing increasing levels of independency.
Change in MoCA | Day 7, 90 and at 65 weeks
  MoCA (Montreal Cognitive Assessment): Score 0-30. Score of 26 or over is considered normal. Lower scores indicates cognitive impairment.
Trail Making Test A | Day 7, 90 and at 65 weeks
  Time in seconds
Trail Making Test B | Day 7, 90 and at 65 weeks
  Time in seconds
Change in forward and backward recall | Day 7, 90 and at 65 weeks
  Test result change over the study period
Change in NEWS score from -4 hours to 0 hours before first tablet to 1,3, 7 days after first capsule | Four hours before the first administration of NR, at administration of the first capsule and 1, 3 an 7 days after administration of first capsule
  NEWS (National Early Warning Score): Score 0-20. High scores indicate high degree of illness.
Change in ECOG status | 14 days prior to admission, baseline, day 7, day 90 and week 65
  Eastern Cooperative Oncology Group (0-5, higher is worse)
Change in GSC | Day 1, 3 and 7
  Glasgow Coma Scale
Change in 4 meter walking test | Baseline, day 7, day 90 and week 65
  Time in seconds
Change in clinical Frailty Score | Baseline, day 7, day 90 and week 65
  Time in seconds
Change in grip strength over three months | Baseline, day 7, day 90 and at 65 weeks
  Kg measured with a handheld dynamometer
Change in CAM-ICU | Baseline and day 1,3,7, and every week of hospitalization in ICU
  CAM-ICU (Confusion Assessment Method for the ICU): Algorithm of Yes/No questions.
Changes in hearing | At baseline, 7 and 90 days and 65 weeks
  Audiogram
Change in left ventricular ejection fraction | Baseline, day 7 and at 90 days
  Measured with echocardiography
Mitochondrial biogenesis - Respiratory Chain Enzyme Analysis | Baseline and 90 days
  Change from baseline in mitochondrial function at the start and end of the 4 weeks of NR treatment (Respiratory chain enzyme analysis)
Change in mitochondrial biogenesis - mitochondrial DNA quantification | Baseline to 90 days
  Change from baseline in the amount of mitochondrial DNA at the start and end of the 90 days of NR treatment (mtDNA quantification)
Change in NAD+ (nicotinamide adenosine dinucleotide) and related metabolite blood levels | Baseline, day 7 and day 90
  Blood samples will be analysed using high performance liquid chromatography-mass spectroscopy and kit-based analysis for levels of NAD+ and related metabolites including: nicotinamide-adenine dinucleotide phosphate, nicotinic acid adenine dinucleotide, nicotinamide, and nicotinamide mononucleotide.
Number of readmissions to hospital | Up to 90 days
  Number
Safety - change in blood analytes | Up to 90 days
  Change from baseline in safety blood analyte levels - Sodium potassium phosphate urea creatinine albumin bilirubin carbamide CRP ALP AST ALT LT GT amylase Mg ferritin hemoglobin leucocytes with subgroups thrombocytes Ca INR PH(venous) HCO3(venous) ProBNP HbA1c TSH fT4 folate homocysteine cholesterol LDL HDL CKMB TNT
Safety - adverse events | Up to 90 days
  Adverse events classified according to CTCAE

OTHER OUTCOMES:
Subgroup analysis - gender | Ut to 90 days
  The primary outcome will be analyzed stratified by gender
Subgroup analysis - age | Ut to 90 days
  The correlation between age and the primary outcome will be measured.
Subgroup analysis - epigenetic age | Ut to 90 days
  The correlation between biological age measured by the DNA methylation based method "GrimAge" (Steve Horvath, 2019 and the primary outcome will be measured.
Subgroup analysis - CRP | Ut to 90 days
  The primary outcome will be analyzed stratified by the maximum measured value of C-reactive protein in plasma of the patient during the hospitalization.
Subgroup analysis - aminoglycosides | Ut to 90 days
  Changes in hearing over the study period will be measured with an audiometer stratified analyses based on the administration of aminoglycosides will be conducted.
Subgroup analysis - NR doses | Ut to 90 days
  The primary outcome will be analyzed stratified by NR dose given to participants.
Subgroup analysis - NR doses | Baseline, day 7, day 90 and at 65 weeks
  Grip strength measured in kg with a handheld dynamometer
Subgroup analysis - NR doses | Day 7, 90 and at 65 weeks
  MoCA will be analyzed stratified by NR dose: MoCA (Montreal Cognitive Assessment): Score 0-30. Score of 26 or over is considered normal. Lower scores indicates cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Søraas, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
Sharing of data will be restricted due to European General Data Protection Regulations (GDPR), but the study team will collaborate on analyzing data within these regulations.

DOCUMENTS (2):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT04110028/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT04110028/SAP_001.pdf